CLINICAL TRIAL: NCT02999893
Title: A phase1b/2 Study Evaluating the Efficacy of APR-246, a First-in-class Agent Targeting Mutant p53 in the Treatment of Platinum Resistant Advanced and Metastatic Oesophageal or Gastro-oesophageal Junction Cancers
Brief Title: A Study of APR-246 in Oesophageal Cancer
Acronym: APROC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding ceased
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/012
Record Dates: First submitted 2016-12-05; First posted 2016-12-21 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Oesophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — eprenetapopt

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APR-246 (Experimental): The trial regimen consists of the investigational agent APR-246, along with standard chemotherapy, Cisplatin and 5-FU. A maximum of 8 cycles of treatment will be given.
  APR-246 and 5-FU must both commence on Day 1 and given on days 1 to 4 via intravenous infusion over 6 hours, whilst 5-FU must be given as a continuous infusion over 96 hours.
  On Days 2-4, APR-246 must be given first via intravenous infusion over 6 hours, then commence cisplatin via intravenous infusion over one hour.
  This is a dose-escalation study to determine the maximum tolerated dose (MTD) of the combination therapy. The 3 dose levels are described as follows:
  Dose Level 1:
  APR-246 Dose: 75mg/kg LBM Cisplatin Dose: 25mg/m2 5-FU Dose: 750mg/m2/ day CI
  Dose Level 2:
  APR-246 Dose: 100mg/kg LBM Cisplatin Dose: 25mg/m2 5-FU Dose: 750mg/m2/ day CI
  Dose Level -1:
  APR-246 Dose: 50mg/kg LBM Cisplatin Dose: 25mg/m2 5-FU Dose: 750mg/m2/ day CI
  Interventions: Drug: APR-246

INTERVENTIONS:
Drug: APR-246 — APR-246 (also known as PRIMA-1MET), a first-in-class agent targeting mutant p53 resulting in re-expression of wild-type p53 activity.

SUMMARY:
The purpose of this study is to determine whether APR-246, 5-FU and cisplatin are safe and effective in the treatment of platinum resistant oesophageal cancer.

DETAILED DESCRIPTION:
Cancer of the oesophagus (OC) is distinguished by having a poor outcome for most patients and an incidence that is rising faster than any other solid cancer. It is already the eighth most common cancer, and the sixth most common cause of death from cancer, worldwide. The majority of patients are diagnosed with late stage disease, which is incurable with the current standard multimodality therapy. Thus, there is a critical need to develop new treatments for this disease.

Surprisingly, despite its high prevalence in developing countries, and its increasing incidence in Western populations, metastatic OC remains an 'orphan disease' with very few good quality or randomised trials available to guide practice. As a result, treatment for OC has changed little over the past few decades, and as a consequence there has been only modest improvement in overall survival for patients with this disease.

TP53, a key tumour suppressor gene, is mutated in 70-80% of OC (both adenocarcinoma and squamous cell carcinoma) providing an attractive potential target for an OC therapy.

Although paired tissue studies in primary and metastatic OC are lacking, p53 mutations occur very early in oesophageal carcinogenesis and are unlikely to be lost in advanced disease. OC with mutant (mut)-p53 are more resistant to conventional chemotherapy and mut-p53 is associated with poor patient prognosis. Over the last decade, several novel drugs have been developed that target mut-p53 and restore wild-type (wt)-p53 function in cancer cells. Of these, APR-246 (also known as PRIMA-1MET), a first-in-class agent targeting mutant p53 resulting in re-expression of wild-type p53 activity, has proven to be the most effective against a wide range of mutants. APR-246 is a pro-drug that gives rise to the active compound methylene quinuclidinone (MQ), which covalently binds to thiol groups on cysteine residues in the p53 core domain resulting in refolding of mut-p53 protein and restoration of its tumour suppressor activity.

While the reactivation of mut-p53 is thought to be the primary mode of action of APR-246, preclinical studies have suggested potential alternative mechanisms (e.g. through the depletion of cellular glutathione levels) may also be contributing to the efficacy of APR-246, especially when used in combination with cisplatin/5-FU chemotherapy. Thus, the anti-tumour activity of APR-246 may not be limited to mut-p53 bearing tumours.

Mutation of p53 is the most common genetic aberration in oesophageal cancer being detected in up to 80% of both oesophageal squamous cell cancers and adenocarcinomas.

APR-246 is a first-in-class agent targeting mutant p53. In vitro and in vivo preclinical models have demonstrated that APR-246 has excellent efficacy in OC (both adenocarcinoma and squamous cell carcinoma) and potently synergises with chemotherapies used in the treatment of OC, restoring sensitivity to chemotherapy-resistant tumours. An initial phase I clinical trial has shown APR-246 to be safe in humans and early results from a currently running phase Ib/II trial of APR-246 with carboplatin and liposomal doxorubicin in ovarian cancer have been promising. Together, these data provide a strong rationale for investigating the efficacy of APR-246 in OC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older at screening
2. Histologically-confirmed metastatic or advanced oesophageal or oesophago-gastric junction adenocarcinoma or squamous cell carcinoma
3. Radiologic disease progression at or within 6 months of platinum containing chemotherapy in the advanced/metastatic or adjuvant setting
4. Measurable disease as per RECIST1.1 criteria
5. Measurable lesions must not have previously had radiotherapy or must have progressed following radiotherapy
6. Patients may have had up to 2 lines of previous chemotherapy in the metastatic/advanced setting or 3 lines including adjuvant therapy. If patients have a maintenance strategy following platinum containing chemotherapy (e.g. fluoropyrimidine alone) this will not be considered a separate line of treatment.
7. Patient has provided written informed consent for the trial
8. Tumour tissue available from the initial surgical resection or any previous biopsies taken at any time before screening. Either a FFPE block or 15 unstained sections from the tumour tissue block must be available for the purpose of translation research studies. Obtaining archived tumour material or unstained sections from an archived tumour block will suffice to meet this requirement. The availability of the tumour material must be confirmed at Screening for a patient to be eligible. If no archival tissue block is available and/or fewer than 15 unstained sections are available, eligibility must be confirmed with the Coordinating Principal Investigator or delegate.
9. Patients must have adequate haematological, renal, hepatic and pulmonary functions as defined by:

   * Absolute neutrophil count ≥1.5 x 109/L
   * Haemoglobin ≥ 10 g/L
   * Platelet count ≥100 x 109/L
   * Total serum bilirubin ≤ 1.5 x upper normal limit
   * Alanine aminotransferase (ALT) ≤ 2.5 x upper normal limit or ≤ 5 x upper limit of normal if liver metastases are present
   * Renal: A creatinine clearance rate of greater than 60 mL/minute
10. Have a performance status of 0 or 1 on the ECOG Performance Scale
11. Life expectancy greater than 3 months
12. Female patients of childbearing potential must be willing to use two methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 60 days after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
13. Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 60 days after the last dose of study therapy.
14. Willing to comply with trial therapy and trial-related investigations and evaluations
15. Willing to consent to the use of their collected tumour specimen and blood samples as detailed in the protocol for future scientific research including but not limited to DNA, RNA and protein based biomarker detection
16. Patient is available for follow up throughout time on trial
17. Recovered from previous toxicities (except alopecia)

Exclusion Criteria:

1. Women who are pregnant or lactating
2. More than 2 lines of previous chemotherapy in the advanced or metastatic setting
3. Previous radiotherapy to all sites of measurable disease without post-radiotherapy progression
4. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the date of registration
5. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
6. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
7. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study
8. Surgery or over 40Gy radiation to the primary tumour within 6 weeks of date of registration
9. Presence of symptomatic or uncontrolled brain or central nervous system metastases which require radiotherapy, surgery or ongoing use of corticosteroids
10. Known HIV positive status, active hepatitis B or C
11. Patients requiring or undergoing concurrent treatment with live vaccines
12. Patients requiring or undergoing concurrent treatment with phenytoin
13. Concurrent malignancy requiring therapy (excluding non-invasive carcinoma or carcinoma in-situ)
14. Common Terminology Criteria for Adverse Events of at least grade 2 neuropathy
15. Patient has hearing loss requiring a hearing aid or intervention indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-02-07 (Actual)

PRIMARY OUTCOMES:
Establish the safety profile of combined APR-246 plus cisplatin and 5FU as measured by the satisfactorily low rate of adverse events described according to NCI CTCAE v 4.03. | 3 weeks post commencement of treatment.

SECONDARY OUTCOMES:
Evidence of clinical efficacy of a combined APR-246 and cisplatin/5FU chemotherapy regimen as confirmed by CT/PET/MRI scan. | 6 and 12 weeks post commencement of treatment.

OTHER OUTCOMES:
Number of patients who will benefit from APR-246 therapy as assessed by quantitation of ctDNA levels in patient serum and plasma samples. | Through study completion, an average of 7 years.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Lipton, MB.BS FRACP, Study Chair — Peter MacCallum Cancer Center
Locations (5):
- Australia (5):
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sunshine Hospital Western Health, Sunshine, Victoria